CLINICAL TRIAL: NCT01345292
Title: Assessment of a Potassium Oxalate-Containing Formulation for the Relief of Dentinal Hypersensitivity
Brief Title: A Study of the Relief of Tooth Sensitivity of an Experimental Mouthrinse Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: KOXDHY0005
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 12027-027 (Experimental): Rinse with 10 ml of the assigned mouthwash for 60 seconds after you brush in your usual manner twice daily for one minute using at least a one-inch strip of the assigned toothpaste
  Interventions: Device: Mouthwash
- 310158077046 (Active Comparator): Brush in your usual manner twice daily for at least one minute using at least a one-inch strip of the assigned toothpaste
  Interventions: Drug: Potassium nitrate toothpaste
- 037000003212 (Placebo Comparator): Brush in your usual manner twice daily for at least one minute using at least a one-inch strip of the assigned toothpaste
  Interventions: Drug: Sodium fluoride toothpaste

INTERVENTIONS:
Device: Mouthwash — Rinse with 10 ml of the assigned mouthwash for 60 seconds after you brush in your usual manner twice daily for one minute using at least a one-inch strip of the assigned toothpaste
  Other Names: 1.40% potassium oxalate sensitive mouthwash
  Arms: 12027-027
Drug: Potassium nitrate toothpaste — Brush in your usual manner twice daily for at least one minute using at least a one-inch strip of the assigned toothpaste
  Other Names: 5% Potassium nitrate toothpaste; Sensodyne Original
  Arms: 310158077046
Drug: Sodium fluoride toothpaste — Brush in your usual manner twice daily for at least one minute using at least a one-inch strip of the assigned toothpaste
  Other Names: Crest Cavity Protection
  Arms: 037000003212

SUMMARY:
This study is for people with sensitive teeth and involves going to the dentist for 4 visits over 6 weeks.

During the first 2 weeks, you will just brush your teeth two times a day with the fluoride toothpaste provided.

Then you will be assigned to a group if you qualify to continue in the study. All groups will get a marketed toothpaste and one group will also get a mouthwash with an experimental ingredient. You will have an equal chance of being assigned to any one of the three groups.

For the next 4 weeks, you will brush with your assigned toothpaste and rinse with your assigned mouthwash if assigned to the mouthwash group. A dentist will look at your mouth, teeth, tongue and gums and check for sensitive teeth. The investigators will see if the mouthwash helps to reduce tooth sensitivity during the study.

DETAILED DESCRIPTION:
This is an observer-blind, randomized, parallel-group, single-center, controlled clinical trial. Approximately 246 generally healthy adults meeting the necessary inclusion/exclusion criteria will be enrolled so that 210 subjects (70 per group) would reasonably be expected to complete the study. Subjects will have their oral soft/hard tissues assessed and will be evaluated for sensitivity levels at Screening (Visit 1), Baseline (Visit 2), Visit 3 at Week 2 and Visit 4 at Week 4. During the first two weeks of the study, subjects will be instructed to brush their teeth for one minute in their usual manner, twice daily, using the provided standard fluoride toothpaste. Subjects will return for the Baseline exam and, upon qualification with entry criteria, will be assigned to one of three treatment groups. Qualified subjects will be instructed to brush their teeth two times daily for one minute in their usual manner using the provided toothpaste (standard fluoride toothpaste or 5% potassium nitrate toothpaste). Subjects assigned to the mouthrinse group will be instructed to rinse twice daily, after brushing, with the provided mouthrinse for 60 seconds using 10 ml, for 4 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years of age in good general and oral health without any known allergy to commercial dental products or cosmetics.
* Evidence of a personally signed and dated informed consent document indicating the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial.
* Willingness to use the assigned products according to instructions, availability for appointments, and likelihood of completing the clinical trial.
* The appropriate number and location of eligible teeth, based on protocol-defined standards.
* Adequate oral hygiene (i.e., brush teeth daily and exhibit no signs of oral neglect).

Exclusion Criteria:

* Any medical or dental history or condition, or use of any medication or drug, that per protocol or in the opinion of the investigator might compromise subject comfort or safety, or the analysis of study results.
* Volunteers who have been using any of the following within protocol-defined timeframes:

  * home-care bleaching, whitening products or professional bleaching treatment
  * desensitizing agents whether prescribed or over-the-counter
  * sensitivity toothpastes, mouthwash or oral care products used for the treatment of dentinal hypersensitivity
* Women who are pregnant, nursing or plan to become pregnant during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2011-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lynch, DMD, PhD, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide
Locations (1):
- BioSci Research America, Inc., Las Vegas, Nevada, United States

REFERENCES:
- [Derived] Sharma D, McGuire JA, Gallob JT, Amini P. Randomised clinical efficacy trial of potassium oxalate mouthrinse in relieving dentinal sensitivity. J Dent. 2013 Jul;41 Suppl 4:S40-8. doi: 10.1016/S0300-5712(13)70005-8. PMID 23929644

RESULTS

PARTICIPANT FLOW:
Groups:
- Negative Control (Crest Regular Toothpaste): Crest® Cavity Protection Regular Toothpaste (Brushing Only)
- Positive Control (Sensodyne Toothpaste): Sensodyne® Original Toothpaste (Brushing Only)
- 12027-027 (1.40% Potassium Oxalate Mouth Rinse): Crest® Cavity Protection Regular Toothpaste followed by Investigative 1.40% Potassium Oxalate Mouth Rinse (Brushing followed by Mouth Rinse)
Period: Overall Study
Arm/Group | Negative Control (Crest Regular Toothpaste) | Positive Control (Sensodyne Toothpaste) | 12027-027 (1.40% Potassium Oxalate Mouth Rinse)
Started | 75 | 76 | 75
Completed | 73 | 76 | 74
Not Completed | 2 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Negative Control (Crest Regular Toothpaste) | Positive Control (Sensodyne Toothpaste) | 12027-027 (1.40% Potassium Oxalate Mouth Rinse) | Total
Number analyzed (Participants) | 75 | 76 | 75 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (10.65) | 35.8 (12.14) | 37.4 (11.10) | 36.3 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 52 | 50 | 153
  Male | 24 | 24 | 25 | 73
Region of Enrollment [Number; unit: participants]
  USA | 75 | 76 | 75 | 226

OUTCOME MEASURES:

1. Primary Outcome: Mean Tactile Sensitivity Score at Week 4
Description: Tooth sensitivity was measured using a Yeaple probe. The force at which discomfort was felt by the participant was recorded on a scale of 10-80 grams. The score for each participant was calculated by averaging the scores for all study teeth for that participant.
Time Frame: 4 weeks
Population: Analysis was based on the Intent-to-Treat (ITT) analysis set, defined as all randomized participants who used at least one dose of the study product and had baseline and at least one post-baseline efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: grams of force
Arm/Group | Negative Control (Crest Regular Toothpaste) | Positive Control (Sensodyne Toothpaste) | 12027-027 (1.40% Potassium Oxalate Mouth Rinse)
Number analyzed (Participants) | 73 | 76 | 74
grams of force | 10.39 (1.111) | 21.83 (1.086) | 18.72 (1.101)
Statistical Analysis 1: Comparison: Negative Control (Crest Regular Toothpaste) vs Positive Control (Sensodyne Toothpaste); The null hypothesis was no difference in mean outcome between treatment groups. The alternative hypothesis was a difference in mean outcome between treatment groups; Test type: Superiority or Other; p < 0.001, ANCOVA — If Sensodyne is better than Crest Regular (p<0.05), testing would proceed to comparison of Wk 2 Mean Tactile Sensitivity Scores between Sensodyne and Crest Regular. Family-wise error was controlled at 0.05; Terms included treatment and baseline mean tactile sensitivity (Yeaple probe) score; Mean Difference (Final Values) = 11.44, 95% CI 2-sided [8.37 to 14.50], Standard Error of Mean 1.556
Statistical Analysis 2: Comparison: Negative Control (Crest Regular Toothpaste) vs 12027-027 (1.40% Potassium Oxalate Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — If Potassium Oxalate Mouth Rinse is better than Crest Regular (p<0.05), testing would proceed to comparison of Wk 2 Mean Tactile Sensitivity Scores between Potassium Oxalate Mouth Rinse and Crest Regular. Family-wise error was controlled at 0.05; Terms included treatment and baseline mean tactile sensitivity (Yeaple probe) score; Mean Difference (Final Values) = 8.33, 95% CI 2-sided [5.24 to 11.42], Standard Error of Mean 1.566

2. Primary Outcome: Mean Tactile Sensitivity Score at Week 2
Description: as for outcome 1
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: grams of force
Arm/Group | Negative Control (Crest Regular Toothpaste) | Positive Control (Sensodyne Toothpaste) | 12027-027 (1.40% Potassium Oxalate Mouth Rinse)
Number analyzed (Participants) | 75 | 76 | 74
grams of force | 10.10 (0.576) | 13.16 (0.571) | 12.51 (0.579)
Statistical Analysis 1: Comparison: Negative Control (Crest Regular Toothpaste) vs Positive Control (Sensodyne Toothpaste); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided). Family-wise error was controlled at 0.05; Terms included treatment and baseline mean tactile sensitivity (Yeaple probe) score; Mean Difference (Final Values) = 3.05, 95% CI 2-sided [1.45 to 4.65], Standard Error of Mean 0.812
Statistical Analysis 2: Comparison: Negative Control (Crest Regular Toothpaste) vs 12027-027 (1.40% Potassium Oxalate Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.004, ANCOVA — The significance threshold level was 0.05 (two-sided). Family-wise error was controlled at 0.05; Terms included treatment and baseline mean tactile sensitivity (Yeaple probe) score; Mean Difference (Final Values) = 2.41, 95% CI 2-sided [0.80 to 4.02], Standard Error of Mean 0.818

3. Secondary Outcome: Mean Tactile Sensitivity Visual Analog Scale (VAS) Score at Week 2
Description: Tooth sensitivity was measured using a VAS. At each visit, participants rated their perception of the pain/discomfort experienced from the Yeaple probe by marking a single vertical line on a VAS scale from 0 to 100 mm, where 0 = No Pain/Discomfort and 100 = Intense Pain/Discomfort. The dental recorder measured the length of the line from 0 to the participant's line and recorded the VAS score in mm. The investigator recorded a VAS score of 0 mm for participants who did not experience discomfort at the maximum force of 80 grams. The score for each participant was calculated by averaging the scores for all study teeth for that participant.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | Negative Control (Crest Regular Toothpaste) | Positive Control (Sensodyne Toothpaste) | 12027-027 (1.40% Potassium Oxalate Mouth Rinse)
Number analyzed (Participants) | 75 | 76 | 74
units on a scale (mm) | 41.59 (1.478) | 39.52 (1.471) | 37.16 (1.485)
Statistical Analysis 1: Comparison: Negative Control (Crest Regular Toothpaste) vs Positive Control (Sensodyne Toothpaste); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.324, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean tactile sensitivity VAS score; Mean Difference (Final Values) = -2.06, 95% CI 2-sided [-6.19 to 2.06], Standard Error of Mean 2.091
Statistical Analysis 2: Comparison: Negative Control (Crest Regular Toothpaste) vs 12027-027 (1.40% Potassium Oxalate Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.035, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean tactile sensitivity VAS score; Mean Difference (Final Values) = -4.43, 95% CI 2-sided [-8.56 to -0.31], Standard Error of Mean 2.093

4. Secondary Outcome: Mean Tactile Sensitivity VAS Score at Week 4
Description: as for outcome 3
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | Negative Control (Crest Regular Toothpaste) | Positive Control (Sensodyne Toothpaste) | 12027-027 (1.40% Potassium Oxalate Mouth Rinse)
Number analyzed (Participants) | 73 | 76 | 74
units on a scale (mm) | 39.49 (1.815) | 30.94 (1.782) | 29.32 (1.799)
Statistical Analysis 1: Comparison: Negative Control (Crest Regular Toothpaste) vs Positive Control (Sensodyne Toothpaste); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean tactile sensitivity VAS score; Mean Difference (Final Values) = -8.55, 95% CI 2-sided [-13.6 to -3.52], Standard Error of Mean 2.551
Statistical Analysis 2: Comparison: Negative Control (Crest Regular Toothpaste) vs 12027-027 (1.40% Potassium Oxalate Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean tactile sensitivity VAS score; Mean Difference (Final Values) = -10.2, 95% CI 2-sided [-15.2 to -5.13], Standard Error of Mean 2.553

5. Secondary Outcome: Mean Cold Air Stimulus VAS Score at Week 2
Description: Tooth sensitivity was measured using a Cold Air Stimulus. When being assessed, participants rated their perception of the pain/discomfort experienced when cold air was directed at the exposed root of each tooth by marking a single vertical line on a VAS scale from 0 to 100 mm, where 0 = No Pain/Discomfort and 100 = Intense Pain/Discomfort. The dental recorder measured the length of the line from 0 to the participant's line and recorded the VAS score in mm. The score for each participant was calculated by averaging the scores for all study teeth for that participant.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | Negative Control (Crest Regular Toothpaste) | Positive Control (Sensodyne Toothpaste) | 12027-027 (1.40% Potassium Oxalate Mouth Rinse)
Number analyzed (Participants) | 75 | 76 | 74
units on a scale (mm) | 43.65 (1.612) | 38.74 (1.600) | 40.22 (1.623)
Statistical Analysis 1: Comparison: Negative Control (Crest Regular Toothpaste) vs Positive Control (Sensodyne Toothpaste); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.032, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean cold air stimulus VAS score; Mean Difference (Final Values) = -4.91, 95% CI 2-sided [-9.38 to -0.43], Standard Error of Mean 2.271
Statistical Analysis 2: Comparison: Negative Control (Crest Regular Toothpaste) vs 12027-027 (1.40% Potassium Oxalate Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.136, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean cold air stimulus VAS score; Mean Difference (Final Values) = -3.42, 95% CI 2-sided [-7.93 to 1.09], Standard Error of Mean 2.288

6. Secondary Outcome: Mean Cold Air Stimulus VAS Score at Week 4
Description: as for outcome 5
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | Negative Control (Crest Regular Toothpaste) | Positive Control (Sensodyne Toothpaste) | 12027-027 (1.40% Potassium Oxalate Mouth Rinse)
Number analyzed (Participants) | 73 | 76 | 74
units on a scale (mm) | 39.54 (1.792) | 28.36 (1.755) | 29.30 (1.780)
Statistical Analysis 1: Comparison: Negative Control (Crest Regular Toothpaste) vs Positive Control (Sensodyne Toothpaste); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean cold air stimulus VAS score; Mean Difference (Final Values) = -11.2, 95% CI 2-sided [-16.1 to -6.23], Standard Error of Mean 2.508
Statistical Analysis 2: Comparison: Negative Control (Crest Regular Toothpaste) vs 12027-027 (1.40% Potassium Oxalate Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean cold air stimulus VAS score; Mean Difference (Final Values) = -10.2, 95% CI 2-sided [-15.2 to -5.25], Standard Error of Mean 2.527

7. Secondary Outcome: Global Subjective VAS Score at Week 2
Description: At each visit, participants rated their perception of the pain/discomfort experienced by marking a single vertical line on a VAS scale from 0 to 100 mm, where 0 = No Pain/Discomfort and 100 = Intense Pain/Discomfort. Participants were instructed as follows: "Please rate the intensity of the pain/discomfort you have experienced in the last two weeks when drinking cold/hot beverages and/or foods, eating sweet and sour foods, breathing cold air, brushing your teeth or performing any habits/behaviors that solicit your dentinal hypersensitivity pain/discomfort since you first started using the product." The dental recorder measured the length of the line from 0 to the participant's line and recorded the VAS score in mm.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | Negative Control (Crest Regular Toothpaste) | Positive Control (Sensodyne Toothpaste) | 12027-027 (1.40% Potassium Oxalate Mouth Rinse)
Number analyzed (Participants) | 75 | 76 | 74
units on a scale (mm) | 44.94 (1.426) | 43.68 (1.416) | 43.64 (1.434)
Statistical Analysis 1: Comparison: Negative Control (Crest Regular Toothpaste) vs Positive Control (Sensodyne Toothpaste); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.533, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean global subjective VAS score; Mean Difference (Final Values) = -1.26, 95% CI 2-sided [-5.22 to 2.71], Standard Error of Mean 2.012
Statistical Analysis 2: Comparison: Negative Control (Crest Regular Toothpaste) vs 12027-027 (1.40% Potassium Oxalate Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.522, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean global subjective VAS score; Mean Difference (Final Values) = -1.30, 95% CI 2-sided [-5.29 to 2.69], Standard Error of Mean 2.023

8. Secondary Outcome: Global Subjective VAS Score at Week 4
Description: as for outcome 7
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | Negative Control (Crest Regular Toothpaste) | Positive Control (Sensodyne Toothpaste) | 12027-027 (1.40% Potassium Oxalate Mouth Rinse)
Number analyzed (Participants) | 73 | 76 | 74
units on a scale (mm) | 41.32 (1.664) | 32.79 (1.630) | 35.19 (1.651)
Statistical Analysis 1: Comparison: Negative Control (Crest Regular Toothpaste) vs Positive Control (Sensodyne Toothpaste); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean global subjective VAS score; Mean Difference (Final Values) = -8.53, 95% CI 2-sided [-13.1 to -3.94], Standard Error of Mean 2.331
Statistical Analysis 2: Comparison: Negative Control (Crest Regular Toothpaste) vs 12027-027 (1.40% Potassium Oxalate Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.010, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean global subjective VAS score; Mean Difference (Final Values) = -6.13, 95% CI 2-sided [-10.8 to -1.51], Standard Error of Mean 2.344

ADVERSE EVENTS:
Time Frame: Day 28 ±3 days, +30 days for serious adverse events.
Description: Adverse events were systematically collected at each study visit through Visit 4 (Day 28 ±3 days). Serious adverse events were reported through 30 days after product use. Spontaneously reported adverse events collected outside of the regularly scheduled visits were also recorded.
Arm/Group | Negative Control (Crest Regular Toothpaste) | Positive Control (Sensodyne Toothpaste) | 12027-027 (1.40% Potassium Oxalate Mouth Rinse)
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/76 | 0/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/76 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigator agreed not to publish the study results without prior sponsor approval.